CLINICAL TRIAL: NCT04462653
Title: Evaluation of the Consistency Between the Detection of Atrial Fibrillation by a Wearable Dynamic ECG Recorder and a Control Instrument
Brief Title: Evaluation of the Detection of Atrial Fibrillation by a Wearable Dynamic ECG Recorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huami Corporation (Industry)
Responsible Party: Principal Investigator, Ruogu.li, Chief Physician, Shanghai Chest Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: BZYL-5-1
Record Dates: First submitted 2020-05-06; First posted 2020-07-08 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- use two kinds of device successively (Experimental): the same participant use a Wearable Dynamic ECG Recorder and 12-lead ECG to record heart rate and atrial fibrillation
  Interventions: Device: Wearable Dynamic ECG Recorder; Device: 12-lead ECG recordings

INTERVENTIONS:
Device: Wearable Dynamic ECG Recorder — use a Wearable Dynamic ECG Recorder to record heart rate and atrial fibrillation
Device: 12-lead ECG recordings — use a 12-lead ECG recordings to record heart rate and atrial fibrillation

SUMMARY:
A Randomized, Crossover Trial is conducted to Evaluate Consistency Atrial fibrillation diagnosis between the Wearable Dynamic ECG Recorder and the Control device.

In this investigation, the following indicators is also evaluated:

1. Sensitivity and specificity of the ECG App algorithm in detecting atrial fibrillation compared with physician-adjudicated Gold Standard ECG recorder.
2. Waveform qualitative assessment
3. Safety incident assessments. 114 subjects (60 healthy subjects in phase I and 54 subjects with atrial fibrillation diagnosis in phase II) are enrolled in the investigation according to the criteria.

ELIGIBILITY:
Inclusion Criteria:

* - All study participants must be able to provide written informed consent prior to study procedure. This study has 2 Phases.

Phase 1:

* Health conscious individuals
* > 18 years of age

Phase 2:

* > 18 years of age
* non critical patients ever diagnosed with atrial fibrillation

Exclusion Criteria:

* • < 18 years old

  * Unable to consent

Phase 1:

* > 80 years of age
* Previous history of cardiac disease (e.g., atrial fibrillation, myocardial infarction, congestive heart failure)
* current status of non-sinus heart rhythm

Phase 2:

- Critical patients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2020-04-24 (Actual); Primary Completion 2020-08-01 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
Consistent rate of atrial fibrillation diagnosis | second 60
  Electrical signals from ECG electrodes are collected with tested device and gold standard device. An automatic diagnosis of atrial fibrillation made with the tested device, and diagnosis of atrial fibrillation is made by the investigators with gold standard device. Diagnosis results include: "with atrial fibrillation (AF)", "without atrial fibrillation (No AF)", or "indecipherable".
  After the diagnosis, the number of "with atrial fibrillation (AF)", "without atrial fibrillation (No AF)", or "indecipherable" cases measured by the two devices are calculated according to table 1, and then the results are evaluated for 3×3 matching consistency.

SECONDARY OUTCOMES:
Sensitivity and specificity of the ECG App algorithm in detecting atrial fibrillation | second 60
  Sensitivity and specificity of the ECG App algorithm in detecting atrial fibrillation compared with physician-adjudicated Gold Standard ECG recorder. Per the protocol, only readable and classifiable (classifiable analysis set) paired recordings are included in the diagnostic performance assessment.
waveform qualitative assessment 1 | second 60
  1)The proportion of paired ECG strips appear to overlay to the unaided eye > 0.80.
waveform qualitative assessment 2 | second 60
  2)The proportion of paired R-wave amplitude measurements within 2 mm of each other > 0.80

OTHER OUTCOMES:
Safety measures 1 | second 60
  1.Scoring system for skin reaction:No erythema, score 0; Very slight erythema (barely perceptible), score 1; Well-defined erythema, score2;Moderate erythema, score 3;Severe erythema (beet-redness) to eschar formation preventing grading of erythema, score 4.
Safety measures 2 | second 60
  2. Adverse event (AE)
Safety measures 3 | second 60
  3. Equipment defector failure for example: unable to wear, no results output, signal interruption.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest hospital, Shanghai, China